CLINICAL TRIAL: NCT03941028
Title: Clinical Effects of Large Segmental Bone Defects Caused by Trauma, Infection and Tumor With 3D Printed Titanium Implant
Brief Title: Clinical Effects of Large Segmental Bone Defects With 3D Printed Titanium Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Z181100001718195
Record Dates: First submitted 2019-04-15; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Large Segmental Bone Defect

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bone defects caused by trauma (Experimental): Large bone defects (>6cm) caused by trauma
  Interventions: Device: 3D printed titanium implant
- bone defects caused by infection (Experimental): Large bone defects caused by chronic osteomyelitis
  Interventions: Device: 3D printed titanium implant
- bone defects caused by tumor (Experimental): Large bone defects caused by benign tumor
  Interventions: Device: 3D printed titanium implant

INTERVENTIONS:
Device: 3D printed titanium implant — The 3D printed titanium implant is fabricated by related companies. And some implants have been used in spinal disease in our hospital.

SUMMARY:
The investigators apply 3D printed titanium implant to treat bone defects. Without using bone grafts and growth factors, the investigators anticipate the titanium implant alone can help bone reconstruction.

DETAILED DESCRIPTION:
The investigators treat large segmental bone defects caused by three reasons, including trauma, infection and tumor. In this study, polyporous 3D printed titanium implant is applied to reconstruct the bone defects and the investigators will follow up patients' function and bone regeneration.

ELIGIBILITY:
Inclusion Criteria:

* bone defects caused by trauma or infection or tumor
* the length of bone defect is more than 6cm
* more than 18 years old

Exclusion Criteria:

* malignant tumor
* patients with bad conditions failing to tolerate surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-12 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Bone reconstruction | 1 year
  X-rays and CT scans are used to evaluate the bone reconstruction

SECONDARY OUTCOMES:
Questionnaire of limb function | 1 year
  Restoration of limb function.

OTHER OUTCOMES:
Questionnaire of patients' satisfaction degree | 1 year
  VAS score is used to evaluate the satisfaction degree. The score ranges from 0 to 10, 0 means very dissatisfied and 10 means very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Tian, MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No